CLINICAL TRIAL: NCT03348423
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo- and Active-Controlled, Evaluation of the Efficacy and Safety of DEX-IN Following Painful Outpatient Procedures
Brief Title: Evaluation of DEX-IN During Outpatient Procedures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baudax Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC-17-023
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-04

CONDITIONS: Pain
Keywords: Peri-procedural pain; Pain; Anxiety; Analgesia; Anxiolysis
MeSH Terms: conditions — Pain; Anxiety Disorders; Agnosia | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, double-dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DEX-IN 50 µg (Experimental): Dexmedetomidine Intranasal Spray
  Interventions: Drug: DEX-IN
- Fentanyl 50 µg (Active Comparator): Intravenous Fentanyl
  Interventions: Drug: Fentanyl
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DEX-IN — IN Dexmedetomidine + IV placebo
  Arms: DEX-IN 50 µg
Drug: Fentanyl — IN Placebo + IV Fentanyl
  Arms: Fentanyl 50 µg
Drug: Placebo — IN Placebo + IV Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the analgesic efficacy of DEX-IN compared with placebo and active control (fentanyl), in subjects undergoing painful outpatient and office based procedures.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent
* Be planned to undergo a selected office-based or outpatient procedure
* Be naïve to the planned procedure, i.e. no repeated or revision procedures
* Not pregnant or planning to become pregnant, or using appropriate contraceptive measures.

Exclusion Criteria:

* Known allergy to any study treatment or excipient
* Have another painful physical condition or anxiety related diagnosis that may confound study assessments
* Evidence of a clinically significant finding on physical examination, laboratory assessment, or ECG
* Have signs or a history of significant nasal condition that may interfere with intranasal drug delivery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DEX-IN 50 µg | Fentanyl 50 µg | Placebo
Started | 15 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | DEX-IN 50 µg | Fentanyl 50 µg | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (12.76) | 47.2 (9.78) | 46.8 (10.31) | 44.5 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 14 | 40
  Male | 2 | 2 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 12 | 15 | 13 | 40
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Pain Intensity - Mean Pain Score During Procedure
Description: Evaluation of subject reported pain intensity scores according to the 11-point Numeric Pain Rating Scale (NPRS; 0-10)
Time Frame: Up to 4 Hours
Population: Randomized subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DEX-IN 50 µg | Fentanyl 50 µg | Placebo
Number analyzed (Participants) | 15 | 15 | 15
units on a scale | 3.03 (0) | 3.10 (0) | 4.25 (0)

ADVERSE EVENTS:
Time Frame: 7 Days
Arm/Group | DEX-IN 50 µg | Fentanyl 50 µg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 5/15 | 2/15 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEX-IN 50 µg (N=15) | Fentanyl 50 µg (N=15) | Placebo (N=15)
Blood pressure decrease (Investigations) | 3 (4) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Discussion and/or publication of data generated is not permitted without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT03348423/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT03348423/SAP_001.pdf